CLINICAL TRIAL: NCT04615637
Title: Helium 4 Optically Pumped Magnetometers : a New Generation of Sensors for High Speed Functional Brain Imaging
Acronym: NEW MEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0191; 2020-A00634-35 (Registry Identifier: ID RCB)
Record Dates: First submitted 2020-07-08; First posted 2020-11-04 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Normal Subject; Patient With Pharmaco-resistant Epilepsy
Keywords: MEG; OPM; epilepsy; normal brain activity
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensors (Experimental): All subjects will follow the same experimental procedure: a recording using classical MEG followed by a recording in the same condition with the OPM He4 prototype.
  Interventions: Device: MEG recordings

INTERVENTIONS:
Device: MEG recordings — 1. Classical MEG recordings (patient at rest, normal subjects stimulated with visual, motor, somesthesic and auditory stimuli).
  2. MEG recordings with our OPM He4 prototype (patient at rest, normal subjects stimulated with visual, motor, somesthesic and auditory stimuli).

SUMMARY:
Our goal is to perform a first evaluation of the capabilities of a new generation of non-invasive magnetoencephalography sensors (OPM He4) to record brain magnetic activities. The investigator will record 1) normal subjects stimulated with visual, auditory, somesthesic and motor stimuli and 2) epileptic patient. The investigator will compare the signal to noise ratio of the normal or pathological activities between classical MEG sensors and our OPM He4 prototype.

ELIGIBILITY:
Inclusion Criteria:

Volunteers:

* Age 18+
* Right handed
* Medical insurance
* Strongly motivated to participate to the study
* Signed informed consent for the study
* No previous neurology or psychiatric pathologies
* No major cognitive deficit and able to understand the instructions

Patients:

* Age 18+
* Right handed
* Medical insurance
* Strongly motivated to participate to the study
* Signed informed consent for the study
* No previous neurology or psychiatric pathologies (except epilepsy)
* Epilepsy evolving during at least two years
* No major cognitive deficit and able to understand the instructions

Exclusion Criteria:

Volunteers:

* Age < 18 years or > 60

  * previous neurology or psychiatric pathologies
  * Child bearing women
  * Subject having one of the following mettalic parts :

    * (pacemaker, implentable pump, neurosimulator, chochlear implant, auditory prothesis, mettalic prothesis, intracerebral clip, implantable defibrilator, any mettalic parts in the brain or upper part of the body, ventriculoperitoneal valve)
    * Claustrophobia Woman with a positive pregnancy test during the inclusion.

Patients:

Age < 18 years or > 60

* previous neurology or psychiatric pathologies except epilepsy
* Child bearing women
* Subject having one of the following mettalic parts :

  * (pacemaker, implentable pump, neurosimulator, chochlear implant, auditory prothesis, mettalic prothesis, intracerebral clip, implantable defibrilator, any mettalic parts in the brain or upper part of the body, ventriculoperitoneal valve)
  * Claustrophobia Woman with a positive pregnancy test during the inclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Signal to Noise Ratio of the recorded brain activities | 1 month
  Volunteers: The signal to noise ratio of normal brain activity following a stimulus will be computed with respect to the pre-stimulus baseline -100ms to -10 ms.
  Epileptic patient: The signal to noise ratio of abnormal epileptic brain activity will be computed with respect to a 100 ms baseline not containing any abnormal activity.

SECONDARY OUTCOMES:
Signal to Noise Ratio of pre-frontal auditory activity | one month
  evaluate the capacities of MPO to record pre-frontal auditory activities which are not recorded by classical MEG. EEG will be the reference
Signal to Noise Ratio of high frequency epileptic activity | one month.
  evaluate the capacities of our MPO to record high frequency epileptic signal which are not recorded by current generation of MPO
Comfort of the subject during the MPO He4 recordings for epileptic patient through a short verbal questionary | 5 minutes after the end the recording session
  The evaluation will be done verbally through a short questionary. This questionary evaluates the overall comfort of the MPO system with two questions: 1) An evaluation of the overall comfort thanks to a scale with five steps from very uncomfortable to very comfortable and 2) A comparison with the classical MEG system thanks to a 5 steps scale from much less comfortable than the classical MEG system to much more comfortable.
Comfort of the subject during the MPO He4 recordings for volunteers through a short verbal questionary | 5 minutes after the end of each recording session
  The evaluation will be done verbally through a short questionary. This questionary evaluates the overall comfort of the MPO system with two questions: 1) An evaluation of the overall comfort thanks to a scale with five steps from very uncomfortable to very comfortable and 2) A comparison with the classical MEG system thanks to a 5 steps scale from much less comfortable than the classical MEG system to much more comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Julien JUNG, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No